CLINICAL TRIAL: NCT01167907
Title: Evaluation of a Continuous Saphenous Nerve Block to Supplement a Continuous Sciatic Nerve Block for Postoperative Analgesia Following Ankle Surgery
Brief Title: Evaluation of Continuous Saphenous Nerve Block to Supplement a Continuous Sciatic Nerve Block After Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00013823
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Orthopedic Surgery of Lower Extremity
Keywords: ankle; arthrodesis; internal fixation; bi/tri malleolar fracture
MeSH Terms: conditions — Ankylosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 0.2% ropivacaine (Experimental): Patients with evidence of sciatic and saphenous nerve block will be randomized to receive a postoperative continuous infusion of either saline (control) or 0.2% ropivacaine by elastomeric infusion pump at 5ml/h started within 6h of catheter placement.
  Interventions: Device: 0.2% ropivacaine; Drug: saline
- Saline (Placebo Comparator): Patients with evidence of sciatic and saphenous nerve block will be randomized to receive a postoperative continuous infusion of either saline (control) or 0.2% ropivacaine by elastomeric infusion pump at 5ml/h started within 6h of catheter placement.
  Interventions: Drug: saline

INTERVENTIONS:
Device: 0.2% ropivacaine — 0.2% ropivacaine by elastomeric infusion pump at 5ml/h started within 6h of catheter placement
  Other Names: NAROPIN®
  Arms: 0.2% ropivacaine
Drug: saline — saline (control) by elastomeric infusion pump at 5ml/h started within 6h of catheter placement

SUMMARY:
A nerve block catheter is a small tube placed next to a nerve through a needle, and the needle is then removed. Numbing medicine is dripped through the tube to reduce pain sensation from the nerve.

The purpose of this research study is to test whether the placement of a second nerve block catheter, rather than a single injection for the saphenous nerve block will improve pain relief and/or reduce pain medication needed after surgery enough to justify two nerve block catheters.

There are two nerves that carry pain sensations from the ankle, the large (sciatic) nerve and the smaller (saphenous) nerve. Patients undergoing ankle fusion or fracture surgery at Wake Forest University typically have a nerve block catheter placed next to the sciatic nerve to give local anesthetic (numbing medicine) for 24-72 hours. In addition, a single injection of local anesthetic is usually performed to block the saphenous nerve for 12-16 hours postoperatively.

DETAILED DESCRIPTION:
Interventions and Interactions Study participants will be asked to report a preoperative baseline pain score (Numeric Pain Scale (0-10)), and have quadriceps strength measured (see below) prior to any sedation being administered. Patients will undergo placement of a continuous subgluteal sciatic nerve catheter, and dosage with 25ml of 0.25% bupivacaine with epinephrine 1:200,000 and clonidine 25 mcg per usual technique after sedation. A perineural catheter will then be placed for primary saphenous nerve block and postoperative saphenous infusion. This continuous saphenous catheter will be placed using ultrasound guidance (Sonosite Turbo ™, Bothell, WA) (6-13MHz linear probe). The superficial femoral artery will be identified in short axis at approximately the midpoint or distal third of the femur as the artery lies deep to the sartorius muscle in the adductor canal. Using aseptic technique, an 18 gauge tuohy needle will be inserted in-plane from lateral to the transducer and advanced to a position anteromedial to the artery, between sartorius and vastus medialis muscles. Proper positioning will be confirmed by injection of saline, a 20g multiorifice catheter will be inserted 3-4 cm beyond the needle tip and the catheter will be tunneled and taped up the medial surface of the thigh. The catheter will be test dosed with 1.5% lidocaine with 1:200,000epinephrine to confirm position and rule out IV injection. The primary saphenous nerve block will be produced by incremental injection through the catheter of 10ml of 0.25% bupivacaine with epinephrine 1:200,000 and clonidine 15 mcg. Successful saphenous block will be defined as loss of sensation to pinprick in the mid, anteromedial leg measured at 15 and 30 minutes post-block. A 3-point scale will be used to define sensory block: 0=full sensation, 1= touch without sharp sensation, 2=absent sensation.

To determine the effect of saphenous block on quadriceps function, patients will have knee extension muscle strength tested pre-block and 30 min post-block using a Hoggan Health microFET 2 MT Digital Handheld Dynamometer. After placement of both the saphenous and sciatic nerve catheters, patients will receive either neuraxial or general anesthesia for surgical anesthesia at the discretion of the attending anesthesiologist medically directing their primary anesthetic technique.

Patients with evidence of sciatic and saphenous nerve block will be randomized to receive a postoperative continuous infusion of either saline (control) or 0.2% ropivacaine by elastomeric infusion pump at 5ml/h started within 6h of catheter placement. The randomization will occur by sealed envelope provided to the OR Pharmacy (block randomization in blocks of 10) and the OR pharmacy will prepare the 300 ml elastomeric pump with active or control solution. The On-Q C-Bloc™(300ml capacity) (I-Flow corporation) pump will be attached to the saphenous catheter in the PACU, or within 6h of primary block; the catheter will infuse for 60 hours.

The patients, physicians, nurses and investigators will be blinded to treatment group.

The sciatic infusion will be managed per usual practice: postoperatively all patients will receive 0.2% ropivacaine through their sciatic nerve catheter at a basal infusion rate of 10ml/h, . The sciatic pump will be an On-Q™ pump per usual practice. All patients will have oral and IV opioids prescribed while hospitalized, and oral opioids prescribed after hospital discharge. In the event of breakthrough pain, patients will be instructed to adjust the sciatic nerve pump, and/or to take oral opioids for the pain.

While patients are hospitalized, opioid administration and pain scores will be recorded by nursing staff on the patient care record. Side effects including nausea, vomiting, or itching will also be recorded. Patients will be seen on a daily basis while in the hospital by the acute pain service, and adjustment of their sciatic infusion performed if indicated. They will be questioned about sleep quality, pain score, opioid side effects, and sensory function in the sciatic and saphenous distributions. This information will be recorded by the acute pain management team. On postoperative day 1, all patients will again have their quadriceps muscle group strength assessed with the hand-held dynamometer, and the catheter sites will be inspected per standard protocol.

Patients will be generally discharged home with peripheral nerve catheters in place on POD #1, after receiving written and verbal instructions in perineural catheter management. These patients will be called at 24 and 48 hours post discharge to determine rest and incident numeric pain scores, opioid usage, sleep quality (as number of awakenings for pain), and the presence of nausea or vomiting. Patients will be given contact numbers and instructions to call with any questions or concerns per usual practice.

Outcome Measure(s) The primary endpoint of this study will be a reduction of the rest and incident verbal pain scores 48hpost-nerve blockade when the primary saphenous single-shot block is expected to have resolved. Secondary endpoints of reduction of opioid use, nausea and vomiting, sleep disturbance (as number of awakenings), and reduction of quadriceps strength will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* surgery for unilateral ankle arthrodesis
* surgery for open reduction and internal fixation of bi/tri malleolar fracture

Exclusion Criteria:

* coagulation abnormalities
* history of opioid addiction
* current chronic pain therapy with high dsoe opioid
* allergy to study medication
* failure of the sciatic nerve catheter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weller, M.D., Principal Investigator — Wake Forest Univesity Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.2% Ropivacaine: Patients with evidence of sciatic and saphenous nerve block will be administered 0.2% ropivacaine by elastomeric infusion pump at 5ml/h via the saphenous catheter started within 6h of catheter placement in addition to the sciatic catheter infusion of 0.2% ropivacaine at 10mL/hr.
- Saline: Patients with evidence of sciatic and saphenous nerve block will be administered saline by elastomeric infusion pump at 5ml/h via the saphenous catheter started within 6h of catheter placement in addition to the sciatic catheter infusion of 0.2% ropivacaine at 10mL/hr.
Period: Overall Study
Arm/Group | 0.2% Ropivacaine | Saline
Started | 17 | 15
Completed | 15 | 14
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — saphenous catheter dislodged before comp | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2% Ropivacaine | Saline | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (12.4) | 47.9 (16.8) | 49.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Scores
Description: The primary endpoint of this study will be a reduction of the rest and incident verbal pain scores 48hpost-nerve blockade when the primary saphenous single-shot block is expected to have resolved.
  "Verbal Pain Score" is the outcome measure applied by asking patients to rate their level of pain. The commonly used 11-point numerical pain rating, with 0-10 range is defined as the following: Zero (0) is used to rate "no pain" and is the best score Ten (10) is used to rate "the worst pain imaginable" and is the worst score
Time Frame: 48 hours post nerve blockade
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 15 | 14
units on a scale | 4.2 (3.1) | 5.4 (3.2)

2. Secondary Outcome: Opioid Use
Description: Secondary endpoints of reduction of opioid use will be evaluated.
  Outcome will be measured using 24h mg-equivalent oxycodone consumption. - (Units in mg/24h)
Time Frame: 48 hours post nerve blockade
Measure: Mean (Standard Deviation); unit: mg per 24h
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 15 | 14
mg per 24h | 35.1 (45.4) | 33.3 (27.4)

3. Secondary Outcome: Nausea
Description: Secondary endpoints of reduction of nausea will be evaluated.
Time Frame: 48 hours post nerve blockade
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 14 | 14
Participants | 4 | 1

4. Secondary Outcome: Vomiting
Description: Secondary endpoints of reduction of vomiting will be evaluated.
Time Frame: 48 hour post nerve blockade
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 14 | 14
Participants | 2 | 0

5. Secondary Outcome: Sleep Disturbance
Description: Secondary endpoints of reduction of sleep disturbance (as number of awakenings) will be evaluated.
Time Frame: 48 hours post nerve blockade
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 15 | 14
awakenings | 1.3 (1.9) | 1.6 (2.0)

6. Secondary Outcome: Reduction of Quadriceps Strength
Description: Secondary endpoints of reduction of quadriceps strength will be evaluated. To determine the effect of saphenous block on quadriceps function, patients will have knee extension muscle strength using a Hoggan Health microFET 2 MT Digital Handheld Dynamometer.
  Knee Extension: Measuring knee extension was performed with the digital dynamometer placed on the anterior surface of the lower leg proximal to the ankle.
Time Frame: 24 hours post nerve blockade
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | 0.2% Ropivacaine | Saline
Number analyzed (Participants) | 15 | 14
pounds | 48.1 (22.7) | 37.3 (17.6)

ADVERSE EVENTS:
Time Frame: Adverse events monitored for each patient until study completion, as defined as 48h post block placement.
Description: No difference
Arm/Group | 0.2% Ropivacaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-09-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT01167907/Prot_SAP_000.pdf
  • Informed Consent Form (2013-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT01167907/ICF_001.pdf